CLINICAL TRIAL: NCT04965220
Title: A Phase I Clinical Trial Evaluating the Safety, Tolerability, Pharmacokinetics, and Initial Efficacy of HLX208 (BRAF V600E Inhibitor) in Combination With Trametinib in Patients With Advanced Solid Tumors
Brief Title: HLX208 (BRAF V600E Inhibitor) in Combination With Trametinib in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLX208-MEK-001
Record Dates: First submitted 2021-06-09; First posted 2021-07-16 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Solid Tumor
MeSH Terms: interventions — trametinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ATC (Experimental): HLX208 (dose of RP2D) and trametinib 2mg qd ,orally,Continuation of treatment until progression, withdrawal of informed consent, intolerant toxicity (whichever occurs first)
  Interventions: Drug: HLX 208
- Primary brain tumor (Experimental): HLX208 (dose of RP2D) and trametinib 2mg qd ,orally,Continuation of treatment until progression, withdrawal of informed consent, intolerant toxicity (whichever occurs first)
  Interventions: Drug: HLX 208
- CRC(KRAS mutant) (Experimental): HLX208 (dose of RP2D) and trametinib 2mg qd ,orally,Continuation of treatment until progression, withdrawal of informed consent, intolerant toxicity (whichever occurs first)
  Interventions: Drug: HLX 208
- other solid tumor (Experimental): HLX208 (dose of RP2D) and trametinib 2mg qd ,orally,Continuation of treatment until progression, withdrawal of informed consent, intolerant toxicity (whichever occurs first)
  Interventions: Drug: HLX 208

INTERVENTIONS:
Drug: HLX 208 — take orally
  Other Names: trametinib

SUMMARY:
A phase I clinical trial evaluating the safety, tolerability, pharmacokinetics, and initial efficacy of HLX208 (BRAF V600E inhibitor) in combination with trametinib in patients with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

* 18Y≤Age≤75Y
* Good Organ Function
* Expected survival time ≥ 3 months
* Metastatic/recurrent advanced BRAF+ solid tumors that have been diagnosed histologically and have failed standard treatment
* Previous failure to standard treatment, intolerance to standard treatment, absence of standard treatment, or insuitability for standard treatment at this stage.
* ECOG score 0-1;
* Expected survival time of more than 3 months;

Exclusion Criteria:

* Previous treatment with BRAF inhibitors or MEK inhibitors
* Symptomatic brain or meningeal metastases (unless the patient has been on > treatment for 6 months, has no evidence of progress on imaging within 4 weeks prior to initial administration, and tumor-related clinical symptoms are stable).
* Current or former patients with interstitial lung disease;
* Active clinical severe infection;
* A history of other malignancies within two years, except for cured carcinoma in situ of the cervix or basal cell carcinoma of the skin.
* Other anti-tumor treatments, such as chemotherapy, targeted therapy, or radiation therapy (except palliative radiation therapy), may be given during the study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
MTD | from first dose to the end of Cycle 1 (each cycle is 21 days)
  maximum tolerated dose

SECONDARY OUTCOMES:
RP2D | from first dose to the end of Cycle 1 (each cycle is 21 days)
  Recommended dose for phase II clinical trials
Peak Plasma Concentration (Cmax) of HLX208 | from first dose to the beginning of Cycle 4 (each cycle is 21 days)
  pharmacokinetics
ORR | from first dose to the last patient was followed up for 6 month
  The number of patients with CR or PR divided by the total number of treated patients whose disease was measurable at baseline
Area under the plasma concentration versus time curve (AUC)of HLX208 | from first dose to the beginning of Cycle 4 (each cycle is 21 days)
  pharmacokinetics

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol